CLINICAL TRIAL: NCT02967692
Title: A Randomized, Double-blind, Placebo-controlled, Phase III Study Comparing the Combination of PDR001, Dabrafenib and Trametinib Versus Placebo, Dabrafenib and Trametinib in Previously Untreated Patients With Unresectable or Metastatic BRAF V600 Mutant Melanoma
Brief Title: A Study of the Anti-PD1 Antibody PDR001, in Combination With Dabrafenib and Trametinib in Advanced Melanoma
Acronym: COMBI-i
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPDR001F2301; 2016-002794-35 (EudraCT Number)
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Results first posted 2023-07-24 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Melanoma
Keywords: Spartalizumab (PDR001); dabrafenib; trametinib; melanoma; immunotherapy; PD 1 inhibitor; anti PD1; PD-1; anti-PD-1; combination treatment; malignant skin cancer; skin cancer; BRAF V600; unresectable BRAF V600 mutated melanoma; metastatic BRAF V600 mutated melanoma
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — spartalizumab; dabrafenib; trametinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1 and Part 2 are open- label. Part 3 is double-blind and randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Safety run-in Cohort (Experimental): In Part 1, participants are treated at different dose levels to determine the recommended Phase 3 regimen of spartalizumab in combination with dabrafenib and trametinib. The starting dose of spartalizumab is 400 mg Q4W in combination with the approved dose of dabrafenib (150 mg BID) and trametinib (2 mg QD).
  Interventions: Biological: Spartalizumab; Drug: Dabrafenib; Drug: Trametinib
- Part 2: Biomarker cohort (Experimental): In Part 2, participants are treated with spartalizumab 400 mg Q4W in combination with the approved dose of dabrafenib (150 mg BID) and trametinib (2 mg QD).
  Interventions: Biological: Spartalizumab; Drug: Dabrafenib; Drug: Trametinib
- Part 3- Arm 1: Spartalizumab in combination with dabrafenib and trametinib (Experimental): In Part 3, participants are randomized to receive spartalizumab at the RP3R identified in Part 1 (400 mg Q4W) in combination with approved dose of dabrafenib (150 mg BID) and trametinib (2 mg QD)
  Interventions: Biological: Spartalizumab; Drug: Dabrafenib; Drug: Trametinib
- Part 3- Arm 2: Placebo in combination with dabrafenib and trametinib (Placebo Comparator): In Part 3, participants are randomized to receive matching placebo in combination with the approved dose of dabrafenib (150 mg BID) and trametinib (2 mg QD)
  Interventions: Other: Placebo; Drug: Dabrafenib; Drug: Trametinib

INTERVENTIONS:
Biological: Spartalizumab — Spartalizumab powder for solution is used in Part 1 and Part 2, and as concentrate for solution for infusion for Part 3. Spartalizumab is administered via intravenous infusion over 30 minutes once every 4 weeks
  Other Names: PDR001
  Arms: Part 1: Safety run-in Cohort; Part 2: Biomarker cohort; Part 3- Arm 1: Spartalizumab in combination with dabrafenib and trametinib
Other: Placebo — Placebo is administered via intravenous infusion over 30 minutes once every 4 weeks
  Arms: Part 3- Arm 2: Placebo in combination with dabrafenib and trametinib
Drug: Dabrafenib — Dabrafenib 150 mg capsules BID is administered orally for Days 1-28 of a 28-day cycle, in fasting conditions.
Drug: Trametinib — Trametinib 2 mg tablets QD is administered orally for Days 1-28 of a 28-day cycle, in fasting conditions

SUMMARY:
The purpose of this study was to evaluate safety and efficacy of the combination of an anti-PD-1 antibody (PDR001), a BRAF inhibitor (dabrafenib) and a MEK inhibitor (trametinib) in patients with BRAF V600 mutant, unresectable and metastatic melanoma.

DETAILED DESCRIPTION:
This study was designed as a phase III, multi-center study consisting of 3 parts:

* Part 1: Safety run-in part The safety run-in part aimed to determine the recommended regimen of PDR001 in combination with dabrafenib and trametinib for previously untreated patients with BRAF V600 mutant unresectable or metastatic melanoma (stage IIIC/IV). Spartalizumab was administered at a starting dose level (DL1) of 400 mg every 4 weeks (Q4W), along with fixed doses of dabrafenib (150 mg twice daily) and trametinib (2 mg once daily). The RP3R for Part 3 was determined using the Bayesian Logistic Regression Model (BLRM) with escalation with overdose control (EWOC) criteria.
* Part 2: Biomarker cohort Part 2 was run to explore changes in the immune microenvironment and biomarker modulations upon treatment with the combination of dabrafenib, trametinib and PDR001. Part 2 started when the fourth subject in dose level 1 (DL1) of Part 1 completed approximately 4 weeks of study treatment, and fewer than 3 dose-limiting toxicities (DLTs) were observed. Participants in Part 2 received PDR001 (spartalizumab) at a dosage of 400 mg Q4W, in combination with dabrafenib (150 mg BID) and trametinib (2 mg QD).
* Part 3: Double-blind, randomized, placebo-controlled part Part 3 was comparing the efficacy and safety of spartalizumab in combination with dabrafenib and trametinib to placebo in combination with dabrafenib and trametinib. Part 3 was initiated after determining the RP3R for the combination of spartalizumab with dabrafenib and trametinib in Part 1. Subjects were randomized in a 1:1 ratio to receive either the RP3R dose of spartalizumab identified in Part 1 or placebo, along with dabrafenib (150 mg BID) and trametinib (2 mg QD).

For all parts of the study, the treatment continued until the subject experiences any of the following events: disease progression according to RECIST 1.1 as determined by the Investigator, unacceptable toxicity, initiation of a new anti-neoplastic therapy, pregnancy, withdrawal of consent, physician's decision, loss to follow-up, death, or termination of the study by the Sponsor. Safety evaluations are conducted for all subjects for up to 150 days after the last dose of spartalizumab/placebo (safety follow-up period).

Subjects who discontinued study treatment without disease progression as per RECIST 1.1 continued with tumor assessments according to the protocol until documented disease progression, withdrawal of consent, loss to follow-up, or death, regardless of the initiation of new anti-neoplastic therapy (efficacy follow-up period).

Subjects entered the survival follow-up period after completing the safety follow-up period or experiencing disease progression as per RECIST 1.1 or response criteria for immunotherapy, whichever period is longer (survival follow-up period).

ELIGIBILITY:
Inclusion criteria Part 1: Safety run-in

* Histologically confirmed, unresectable or metastatic melanoma with BRAF V600 mutation
* Aspartate transaminase (AST) < 2.5× ULN and Alanine transaminase (ALT) < 2.5× ULN
* Measurable disease according to RECIST 1.1
* ECOG performance status ≤ 1

Part 2: Biomarker cohort

* Histologically confirmed, unresectable or metastatic melanoma with BRAF V600 mutation
* At least two cutaneous or subcutaneous or nodal lesions for tumor sample collection
* Measurable disease according to RECIST 1.1
* ECOG performance status ≤ 2

Part 3: Double-blind, randomized, placebo-controlled part

* Histologically confirmed, unresectable or metastatic melanoma with BRAF V600 mutation
* ECOG performance status ≤ 2
* Measurable disease according to RECIST 1.1

Exclusion Criteria:

Part 1: Safety run-in

* Subjects with uveal or mucosal melanoma
* Any history of CNS metastases
* Prior systemic anti-cancer treatment for unresectable or metastatic melanoma
* Neoadjuvant and/or adjuvant therapy for melanoma completed less than 6 months prior to enrollmen
* Radiation therapy within 4 weeks prior to start of study treatment
* Active autoimmune disease, and/or history of autoimmune disease(s) that required treatment

Parts 2 & 3: Biomarker cohort & double-blind, randomized, placebo-controlled part

* Subjects with uveal or mucosal melanoma
* Prior systemic anti-cancer treatment for unresectable or metastatic melanoma
* Neoadjuvant and/or adjuvant therapy for melanoma completed less than 6 months prior to enrollment
* Radiation therapy within 4 weeks prior to start of study treatment
* Clinically active cerebral melanoma metastasis.
* Active autoimmune disease, and/or history of autoimmune disease(s) that required treatment

Other protocol-defined Inclusion/Exclusion may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2020-08-11 (Actual); Study Completion 2024-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (166):
- United States (12):
  - California Cancer Associates for Research and Excellence, Encinitas, California
  - UC Irvine Medical Center, Orange, California
  - California Pacific Medical Center, San Francisco, California
  - Stanford Cancer Center, Stanford, California
  - University of Kansas Cancer Center, Westwood, Kansas
  - Johns Hopkins U, Lutherville, Maryland
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - NYU Laura and Isaac Perlmutter Cancer Center, New York, New York
  - University of Pittsburgh Med Center, Pittsburgh, Pennsylvania
  - University of Tennessee Medical Ctr, Knoxville, Tennessee
  - Univ of TX MD Anderson Cancer Cntr, Houston, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
- Argentina (3):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Caba
- Australia (5):
  - Novartis Investigative Site, Gateshead, New South Wales
  - Novartis Investigative Site, North Sydney, New South Wales
  - Novartis Investigative Site, Greenslopes, Queensland
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
- Austria (5):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Sankt Pölten
- Novartis Investigative Site, Brussels, Belgium
- Brazil (4):
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Rio de Janeiro
- Bulgaria (2):
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
- Canada (4):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
- Chile (2):
  - Novartis Investigative Site, Temuco, Región de la Araucanía
  - Novartis Investigative Site, Santiago
- Czechia (6):
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Zlín, Czech Republic
  - Novartis Investigative Site, Hradec Králové, CZE
  - Novartis Investigative Site, Ostrava, Poruba
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Prague
- Novartis Investigative Site, Aarhus N, Denmark
- France (26):
  - Novartis Investigative Site, Limoges, Haute Vienne
  - Novartis Investigative Site, Amiens
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Bobigny
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Boulogne-Billancourt
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lorient
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Mulhouse
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
  - Novartis Investigative Site, Villejuif
- Germany (25):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Halle, Saxony-Anhalt
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Stade
  - Novartis Investigative Site, Tübingen
- Novartis Investigative Site, Athens, Greece
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Szeged
- Israel (3):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Ramat Gan
- Italy (16):
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Meldola, FC
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Candiolo, TO
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Napoli
- Japan (5):
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Kyoto University Hospital, Sakyo Ku, Kyoto
  - Osaka International Cancer Institute, Osaka, Osaka
  - Tokyo Metropolitan Komagome Hospital, Bunkyo Ku, Tokyo
  - National Cancer Hospital, Chuo Ku, Tokyo
- Mexico (3):
  - Novartis Investigative Site, León, Guanajuato
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Mexico City, Mexico City
- Netherlands (2):
  - Novartis Investigative Site, Leiden, South Holland
  - Novartis Investigative Site, Amersfroort
- Novartis Investigative Site, Oslo, Norway
- Poland (2):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Warsaw
- Portugal (2):
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Russia (6):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Omsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Samara
- Spain (10):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Jerez de la Frontera, Cadiz
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Las Palmas de Gran Canaria
  - Novartis Investigative Site, Madrid
- Sweden (3):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Stockholm
- Switzerland (2):
  - Novartis Investigative Site, Aarau, Canton of Aargau
  - Novartis Investigative Site, Zurich
- Thailand (2):
  - Novartis Investigative Site, Songkhla, Hat Yai
  - Novartis Investigative Site, Bangkok
- United Kingdom (9):
  - Novartis Investigative Site, Truro, Cornwall
  - Novartis Investigative Site, Guildford, Surrey
  - Novartis Investigative Site, Sutton, Surrey
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Middlesbrough
  - Novartis Investigative Site, Preston
  - Novartis Investigative Site, Rickmansworth Road

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Tawbi HA, Robert C, Brase JC, Gusenleitner D, Gasal E, Garrett J, Savchenko A, Gorgun G, Flaherty KT, Ribas A, Dummer R, Schadendorf D, Long GV, Nathan PD, Ascierto PA. Spartalizumab or placebo in combination with dabrafenib and trametinib in patients with BRAF V600-mutant melanoma: exploratory biomarker analyses from a randomized phase 3 trial (COMBI-i). J Immunother Cancer. 2022 Jun;10(6):e004226. doi: 10.1136/jitc-2021-004226. PMID 35728875
- [Derived] Dummer R, Long GV, Robert C, Tawbi HA, Flaherty KT, Ascierto PA, Nathan PD, Rutkowski P, Leonov O, Dutriaux C, Mandala M, Lorigan P, Ferrucci PF, Grob JJ, Meyer N, Gogas H, Stroyakovskiy D, Arance A, Brase JC, Green S, Haas T, Masood A, Gasal E, Ribas A, Schadendorf D. Randomized Phase III Trial Evaluating Spartalizumab Plus Dabrafenib and Trametinib for BRAF V600-Mutant Unresectable or Metastatic Melanoma. J Clin Oncol. 2022 May 1;40(13):1428-1438. doi: 10.1200/JCO.21.01601. Epub 2022 Jan 14. PMID 35030011
- [Derived] Dummer R, Lebbe C, Atkinson V, Mandala M, Nathan PD, Arance A, Richtig E, Yamazaki N, Robert C, Schadendorf D, Tawbi HA, Ascierto PA, Ribas A, Flaherty KT, Pakhle N, Campbell CD, Gusenleitner D, Masood A, Brase JC, Gasal E, Long GV. Combined PD-1, BRAF and MEK inhibition in advanced BRAF-mutant melanoma: safety run-in and biomarker cohorts of COMBI-i. Nat Med. 2020 Oct;26(10):1557-1563. doi: 10.1038/s41591-020-1082-2. Epub 2020 Oct 5. PMID 33020648

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part 1 and 2 were conducted in 18 centers across 12 countries. Part 3 is conducted in 190 centers across 29 countries
Pre-assignment Details: The screening phase began once written informed consent was provided and ended after 28 days or when subject received the first dose (Part 1 and 2) or was randomized (Part 3), whichever came first.
Groups:
- Part 1- Safety run-in: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD: In Part 1, participants are treated with Spartalizumab (PDR001) 400 mg Q4W in combination with the approved dose of dabrafenib (150 mg BID) and trametinib (2 mg QD).
- Part 2- Biomarker Cohort: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD: In Part 2, participants are treated with Spartalizumab (PDR001) 400 mg Q4W in combination with the approved dose of dabrafenib (150 mg BID) and trametinib (2 mg QD).
- Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD: In Part 3, participants are randomized to receive Spartalizumab (PDR001) at the RP3R identified in Part 1 (400 mg Q4W) in combination with approved dose of dabrafenib (150 mg BID) and trametinib (2 mg QD)
- Part 3- Arm 2: Placebo + Dabrafenib 150 mg BID + Trametinib 2 mg QD: In Part 3, participants are randomized to receive matching placebo in combination with the approved dose of dabrafenib (150 mg BID) and trametinib (2 mg QD)
Period: Overall Study
Arm/Group | Part 1- Safety run-in: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 2- Biomarker Cohort: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 2: Placebo + Dabrafenib 150 mg BID + Trametinib 2 mg QD
Started | 9 | 27 | 267 | 265
Treated | 9 | 27 | 267 | 264
Completed | 0 | 0 | 0 | 0
Not Completed | 9 | 27 | 267 | 265
Not completed — Progressive disease | 3 | 15 | 114 | 151
Not completed — Subject/guardian decision | 1 | 1 | 14 | 22
Not completed — Death | 0 | 1 | 13 | 13
Not completed — Protocol deviation | 1 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 22 | 13
Not completed — Adverse Event | 2 | 9 | 60 | 28
Not completed — Study terminated by sponsor | 2 | 1 | 42 | 37

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1- Safety run-in: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 2- Biomarker Cohort: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 2: Placebo + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Total
Number analyzed (Participants) | 9 | 27 | 267 | 265 | 568
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 18 | 189 | 195 | 409
  >=65 years | 2 | 9 | 78 | 70 | 159
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 12 | 119 | 106 | 239
  Male | 7 | 15 | 148 | 159 | 329
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9 | 24 | 225 | 227 | 485
  Asian | 0 | 2 | 5 | 5 | 12
  Other | 0 | 1 | 15 | 14 | 30
  Unknown | 0 | 0 | 22 | 19 | 41

OUTCOME MEASURES:

1. Primary Outcome: Safety Run-In (Part 1): Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT was defined as an adverse event or abnormal laboratory value that was unrelated to disease, disease progression, inter-current illness, or concomitant medications and occured within 8 weeks of treatment with spartalizumab in combination with dabrafenib and trametinib. The DLT criteria included Grade 4 hematological adverse events, Grade 4 bilirubin elevation, specific gastrointestinal adverse events, symptomatic serum amylase or lipase elevation, Grade 3 or higher hypertension, Grade 3 or higher cardiac events, Grade 2 or higher pneumonitis, Grade 3 or higher immune-related toxicities, infusion-related reactions, other clinically significant adverse events, and toxicities leading to a dosing delay of over 12 weeks. NCI CTCAE v4.03 was used for grading DLTs
Time Frame: Up to 8 weeks (Part 1)
Population: Dose-Determining Set (DDS) including all subjects in Part 1 who received at least one dose of study treatment who either 1) met the minimum exposure criterion and had sufficient safety evaluations, or 2) experienced a DLT during the first 8 weeks (56 days) of spartalizumab in combination with dabrafenib and trametinib dosing.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1- Safety run-in: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD
Number analyzed (Participants) | 9
Participants | 1

2. Primary Outcome: Biomarker Cohort (Part 2): Change From Baseline in Programmed Cell Death-ligand 1 (PD-L1) Expression Upon Treatment With Spartalizumab in Combination With Dabrafenib and Trametinib
Description: Change from baseline in PD-L1 expression (as determined by immunohistochemistry in tissue samples) upon treatment with spartalizumab in combination with dabrafenib and trametinib in participants from Part 2
Time Frame: Baseline, Cycle 1 Day 15 and Cycle 3 Day 1 (Part 2). Each cycle is 28 days
Population: Participants in Part 2 who received at least one dose of study treatment and with evaluable data at the pre-specified time points
Measure: Mean (Standard Deviation); unit: Percentage of positive tumor cells
Arm/Group | Part 2- Biomarker Cohort: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD
Number analyzed (Participants) | 9
Percentage of positive tumor cells
  Cycle 1 Day 15 | 1.7 (13.05)
  Cycle 3 Day 1: number analyzed (Participants) | 7
  Cycle 3 Day 1 | 2.7 (7.63)

3. Primary Outcome: Biomarker Cohort (Part 2): Change From Baseline in CD8+ Cells Upon Treatment With Spartalizumab in Combination With Dabrafenib and Trametinib
Description: Change from baseline in CD8+ cells (as determined by flow cytometry in blood samples) upon treatment with spartalizumab in combination with dabrafenib and trametinib in participants from Part 2
Time Frame: Baseline, Cycle 1 Day 15 and Cycle 3 Day 1 (Part 2). Each cycle is 28 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage Marker Area
Arm/Group | Part 2- Biomarker Cohort: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD
Number analyzed (Participants) | 6
Percentage Marker Area
  Cycle 1 Day 15 | 0.4 (3.22)
  Cycle 3 Day 1: number analyzed (Participants) | 4
  Cycle 3 Day 1 | 1.2 (2.43)

4. Primary Outcome: Randomized (Part 3): Progression-Free Survival (PFS) as Per Investigator's Assessment by RECIST 1.1
Description: Progression-free survival was defined as the time from the date of first dose to the date of the first documented radiological progression per investigator's assessment according to RECIST 1.1 or death due to any cause. The distribution of PFS was estimated using the Kaplan-Meier (KM) method. If a patient had not had an event at the time of data cut-off, progression-free survival was censored at the date of last adequate tumor assessment.
Time Frame: Up to disease progression or death due to any cause, whichever occurs first, assessed up to 2.8 years (Part 3)
Population: All participants in Part 3 to whom study treatment was assigned by randomization regardless of whether or not treatment was administered.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 2: Placebo + Dabrafenib 150 mg BID + Trametinib 2 mg QD
Number analyzed (Participants) | 267 | 265
Months | 16.2 [12.7 to 23.9] | 12.0 [10.2 to 15.4]
Statistical Analysis 1: Comparison: Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD vs Part 3- Arm 2: Placebo + Dabrafenib 150 mg BID + Trametinib 2 mg QD; Test type: Superiority; p = 0.042, Log Rank; Hazard Ratio (HR) = 0.820, 95% CI 2-sided [0.655 to 1.027]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from date of randomization to date of death due to any cause
Time Frame: Up to death due to any cause, assessed up to approximately 7 years
Population: All participants to whom study treatment was assigned by randomization regardless of whether or not treatment was administered.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1- Safety run-in: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 2- Biomarker Cohort: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 2: Placebo + Dabrafenib 150 mg BID + Trametinib 2 mg QD
Number analyzed (Participants) | 9 | 27 | 267 | 265
Months | NA [12.2 to NA] — Not estimable (NA) due to the insufficient number of participants with events | 30.7 [21.3 to 67.4] | 61.5 [41.6 to NA] — Not estimable (NA) due to the insufficient number of participants with events | 41.6 [30.6 to 56.9]

6. Secondary Outcome: Overall Response Rate (ORR) as Per Investigator's Assessment by RECIST 1.1
Description: ORR was defined as the percentage of subjects with confirmed best overall response of complete response (CR) or partial response (PR), as per investigator's assessment by RECIST 1.1. CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to <10 mm PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters
Time Frame: Part 1: Up to 3.3 years. Part 2: Up to 3 years. Part 3: Up to 2.8 years
Population: For Part 1 and 2: all subjects to whom study treatment was assigned and who received at least one dose of any study treatment. For Part 3: all subjects to whom study treatment was assigned by randomization, regardless of whether or not treatment was administered.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 1- Safety run-in: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 2- Biomarker Cohort: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 2: Placebo + Dabrafenib 150 mg BID + Trametinib 2 mg QD
Number analyzed (Participants) | 9 | 27 | 267 | 265
Percentage of participants | 100.0 [66.4 to 100.0] | 70.4 [49.8 to 86.2] | 68.5 [62.6 to 74.1] | 64.2 [58.1 to 69.9]

7. Secondary Outcome: Duration of Response (DOR) as Per Investigator's Assessment by RECIST 1.1
Description: DOR was defined as the time from first documented response of CR or PR to date of first documented progression or death, according to RECIST 1.1 criteria. The distribution of DOR was estimated using the KM method. CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to <10 mm PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters
Time Frame: From first documented response to date of first documented progression or death, up to 3.3 years (Part 1), 3 years (Part 2) and 2.8 years (Part 3)
Population: For Part 1 and 2: all subjects to whom study treatment was assigned and who received at least one dose of any study treatment for whom best overall response was CR or PR. For Part 3: all subjects to whom study treatment was assigned by randomization (regardless of whether or not treatment was administered) for whom best overall response was CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1- Safety run-in: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 2- Biomarker Cohort: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 2: Placebo + Dabrafenib 150 mg BID + Trametinib 2 mg QD
Number analyzed (Participants) | 9 | 19 | 183 | 170
Months | NA [8.3 to NA] — Not estimable (NA) due to the insufficient number of participants with events | 20.0 [9.4 to NA] — Not estimable (NA) due to the insufficient number of participants with events | NA [18.6 to NA] — Not estimable (NA) due to the insufficient number of participants with events | 20.7 [13.0 to NA] — Not estimable (NA) due to the insufficient number of participants with events

8. Secondary Outcome: Disease Control Rate (DCR) as Per Investigator's Assessment by RECIST 1.1
Description: DCR was defined as the percentage of participants with CR or PR or subjects with stable disease (SD) lasting for a duration of at least 24 weeks as per local review according to RECIST 1.1 criteria. CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to <10 mm PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters SD: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease.
Time Frame: Part 1: Up to 3.3 years. Part 2: Up to 3 years. Part 3: Up to 2.8 year
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 1- Safety run-in: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 2- Biomarker Cohort: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 2: Placebo + Dabrafenib 150 mg BID + Trametinib 2 mg QD
Number analyzed (Participants) | 9 | 27 | 267 | 265
Percentage of participants | 100.0 [66.4 to 100.0] | 92.6 [75.7 to 99.1] | 84.3 [79.3 to 88.4] | 86.4 [81.7 to 90.3]

9. Secondary Outcome: Randomized (Part 3): Change From Baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) C30- Global Health Status Scores
Description: The EORTC QLQ-C30 was a 30-item questionnaire that patients complete, consisting of both multi-item scales and single-item measures. It included five functional scales, three symptom scales, six single items, and a Global Health Status/Quality of Life (GHS/QoL) scale. The GHS/QoL scale had seven possible response scores ranging from 1 (very poor) to 7 (excellent), which were averaged and transformed to a 0-100 scale. A higher score on this scale indicated a better quality of life. The change from baseline in GHS/QoL scores was calculated. A positive change from baseline indicated improvement in the patient's quality of life.
Time Frame: From baseline to 60 days post progression, assessed up to 2.8 years (Part 3)
Population: All participants in Part 3 to whom study treatment was assigned by randomization (regardless of whether or not treatment was administered) and with available data at the pre-specified time points
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 2: Placebo + Dabrafenib 150 mg BID + Trametinib 2 mg QD
Number analyzed (Participants) | 175 | 186
Score on a Scale
  Cycle 4 Day 1 | 0.81 (19.300) | 2.20 (24.918)
  Cycle 6 Day 1: number analyzed (Participants) | 157 | 158
  Cycle 6 Day 1 | 1.22 (25.050) | 1.90 (21.197)
  Cycle 8 Day 1: number analyzed (Participants) | 146 | 151
  Cycle 8 Day 1 | 0.00 (24.526) | 0.50 (19.608)
  Cycle 10 Day 1: number analyzed (Participants) | 133 | 125
  Cycle 10 Day 1 | 1.88 (23.088) | 0.27 (18.752)
  Cycle 12 Day 1: number analyzed (Participants) | 110 | 114
  Cycle 12 Day 1 | 0.61 (25.906) | 0.00 (24.541)
  Cycle 14 Day 1: number analyzed (Participants) | 103 | 103
  Cycle 14 Day 1 | 0.65 (23.561) | -0.89 (23.306)
  Cycle 16 Day 1: number analyzed (Participants) | 91 | 90
  Cycle 16 Day 1 | 0.82 (25.186) | 1.76 (24.142)
  Cycle 18 Day 1: number analyzed (Participants) | 90 | 83
  Cycle 18 Day 1 | -0.46 (24.106) | -0.10 (19.193)
  Cycle 20 Day 1: number analyzed (Participants) | 82 | 82
  Cycle 20 Day 1 | 1.93 (21.766) | -1.02 (23.144)
  Cycle 22 Day 1: number analyzed (Participants) | 79 | 80
  Cycle 22 Day 1 | 0.95 (22.047) | 2.29 (21.947)
  Cycle 25 Day 1: number analyzed (Participants) | 63 | 70
  Cycle 25 Day 1 | 3.57 (23.981) | -0.24 (25.497)
  Cycle 28 Day 1: number analyzed (Participants) | 50 | 55
  Cycle 28 Day 1 | 4.50 (19.793) | 1.06 (22.513)
  Cycle 31 Day 1: number analyzed (Participants) | 23 | 26
  Cycle 31 Day 1 | 11.59 (24.967) | 6.73 (21.084)
  Cycle 34 Day 1: number analyzed (Participants) | 2 | 6
  Cycle 34 Day 1 | 16.67 (47.140) | 13.89 (20.184)
  30 days post-progression: number analyzed (Participants) | 23 | 30
  30 days post-progression | -11.59 (24.967) | -7.78 (29.274)
  60 days post-progression: number analyzed (Participants) | 13 | 16
  60 days post-progression | -11.54 (16.506) | -17.19 (24.050)

10. Secondary Outcome: Randomized (Part 3): Change From Baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) C30- Physical Functioning Scale Scores
Description: The EORTC QLQ-C30 was a patient completed 30 item questionnaire that was composed of both multi-item scales and single-item measures. These included five functional scales, three symptom scales, six single items and a global health status/QoL scale. The EORTC QLQ-C30 physical functioning scale measured a patient's ability to carry out daily activities and tasks requiring physical exertion. It consisted of five questions asking patients to rate their level of physical functioning, with response options ranging from 1="not at all" to 4="very much". The scores for each item were summed and transformed to a 0 to 100 scale, with higher scores indicating better physical functioning. The change from baseline in physical functioning scale scores was calculated. A positive change from baseline indicated improvement in physical functioning.
Time Frame: From baseline to 60 days post progression, assessed up to 2.8 years (Part 3)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 2: Placebo + Dabrafenib 150 mg BID + Trametinib 2 mg QD
Number analyzed (Participants) | 175 | 186
Score on a Scale
  Cycle 4 Day 1 | -1.52 (16.243) | -0.70 (17.618)
  Cycle 6 Day 1: number analyzed (Participants) | 158 | 158
  Cycle 6 Day 1 | -2.38 (16.121) | -0.60 (14.824)
  Cycle 8 Day 1: number analyzed (Participants) | 146 | 150
  Cycle 8 Day 1 | -1.29 (18.350) | -0.59 (15.687)
  Cycle 10 Day 1: number analyzed (Participants) | 133 | 126
  Cycle 10 Day 1 | -0.18 (17.985) | -1.11 (13.736)
  Cycle 12 Day 1: number analyzed (Participants) | 110 | 114
  Cycle 12 Day 1 | -1.39 (18.108) | -0.85 (10.652)
  Cycle 14 Day 1: number analyzed (Participants) | 103 | 103
  Cycle 14 Day 1 | -2.42 (16.720) | -2.61 (12.320)
  Cycle 16 Day 1: number analyzed (Participants) | 91 | 90
  Cycle 16 Day 1 | -4.19 (20.301) | -2.24 (13.331)
  Cycle 18 Day 1: number analyzed (Participants) | 90 | 83
  Cycle 18 Day 1 | -3.48 (18.862) | -3.55 (13.474)
  Cycle 20 Day 1: number analyzed (Participants) | 82 | 82
  Cycle 20 Day 1 | -4.07 (15.316) | -1.73 (11.536)
  Cycle 22 Day 1: number analyzed (Participants) | 79 | 80
  Cycle 22 Day 1 | -3.21 (15.538) | -0.85 (11.157)
  Cycle 25 Day 1: number analyzed (Participants) | 64 | 70
  Cycle 25 Day 1 | -1.35 (16.510) | -2.67 (13.158)
  Cycle 28 Day 1: number analyzed (Participants) | 50 | 55
  Cycle 28 Day 1 | -0.80 (13.843) | -2.67 (15.953)
  Cycle 31 Day 1: number analyzed (Participants) | 23 | 26
  Cycle 31 Day 1 | -2.03 (10.719) | -1.79 (9.533)
  Cycle 34 Day 1: number analyzed (Participants) | 3 | 6
  Cycle 34 Day 1 | 0.00 (0.000) | -3.33 (5.578)
  30 days post-progression: number analyzed (Participants) | 23 | 30
  30 days post-progression | -6.67 (18.641) | -8.67 (19.973)
  60 days post-progression: number analyzed (Participants) | 13 | 16
  60 days post-progression | -13.85 (15.977) | -21.25 (27.991)

11. Secondary Outcome: Randomized (Part 3): Change From Baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) C30- Pain Symptom Scale Scores
Description: The EORTC QLQ-C30 was a patient completed 30 item questionnaire that was composed of both multi-item scales and single-item measures. These included five functional scales, three symptom scales, six single items and a global health status/QoL scale. The EORTC QLQ-C30 pain symptom scale was one of the symptom scales in the questionnaire, which measured the severity of pain experienced by the patient. The pain symptom scale consisted of two items, one measuring the severity of pain and the other measuring the use of painkillers. The items were rated on a 4-point scale ranging from 1="not at all" to 4="very much". The scores for each item were summed and transformed to a 0 to 100 scale, with higher scores indicating more severe pain. The change from baseline in pain symptom scale scores was calculated. A negative change from baseline indicated improvement.
Time Frame: From baseline to 60 days post progression, assessed up to 2.8 years (Part 3)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 2: Placebo + Dabrafenib 150 mg BID + Trametinib 2 mg QD
Number analyzed (Participants) | 175 | 186
Score on a Scale
  Cycle 4 Day 1 | -5.24 (26.434) | -5.29 (24.881)
  Cycle 6 Day 1: number analyzed (Participants) | 158 | 158
  Cycle 6 Day 1 | -6.43 (28.820) | -7.49 (23.611)
  Cycle 8 Day 1: number analyzed (Participants) | 146 | 150
  Cycle 8 Day 1 | -4.91 (29.176) | -4.11 (24.420)
  Cycle 10 Day 1: number analyzed (Participants) | 132 | 126
  Cycle 10 Day 1 | -7.95 (28.346) | -4.76 (23.557)
  Cycle 12 Day 1: number analyzed (Participants) | 110 | 114
  Cycle 12 Day 1 | -8.33 (28.890) | -5.26 (22.646)
  Cycle 14 Day 1: number analyzed (Participants) | 103 | 103
  Cycle 14 Day 1 | -5.50 (28.140) | -3.56 (23.062)
  Cycle 16 Day 1: number analyzed (Participants) | 91 | 90
  Cycle 16 Day 1 | -5.86 (26.220) | -4.44 (25.820)
  Cycle 18 Day 1: number analyzed (Participants) | 90 | 83
  Cycle 18 Day 1 | -3.15 (30.178) | -3.21 (20.898)
  Cycle 20 Day 1: number analyzed (Participants) | 82 | 82
  Cycle 20 Day 1 | -4.47 (30.659) | -2.85 (23.249)
  Cycle 22 Day 1: number analyzed (Participants) | 79 | 80
  Cycle 22 Day 1 | -5.49 (27.049) | -3.54 (23.969)
  Cycle 25 Day 1: number analyzed (Participants) | 64 | 70
  Cycle 25 Day 1 | -6.25 (28.868) | -4.76 (20.685)
  Cycle 28 Day 1: number analyzed (Participants) | 50 | 55
  Cycle 28 Day 1 | -3.00 (26.872) | -3.03 (22.701)
  Cycle 31 Day 1: number analyzed (Participants) | 23 | 26
  Cycle 31 Day 1 | -10.14 (24.995) | -7.05 (34.696)
  Cycle 34 Day 1: number analyzed (Participants) | 2 | 6
  Cycle 34 Day 1 | -8.33 (11.785) | -5.56 (8.607)
  30 days post-progression: number analyzed (Participants) | 23 | 30
  30 days post-progression | 9.42 (28.791) | 0.56 (28.190)
  60 days post-progression: number analyzed (Participants) | 13 | 16
  60 days post-progression | 15.38 (19.792) | 11.46 (24.884)

12. Secondary Outcome: Randomized (Part 3): Time to 10 Point Definitive Deterioration in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) C30- Global Health Status
Description: The EORTC QLQ-C30 was a patient completed 30 item questionnaire that was composed of both multi-item scales and single-item measures. These included five functional scales, three symptom scales, six single items and a global health status/QoL scale. The GHS/QoL scale had seven possible response scores ranging from 1 (very poor) to 7 (excellent), which were averaged and transformed to a 0-100 scale. A higher score on this scale indicated a better quality of life. The time to definitive 10 point deterioration is defined as the time from the date of randomization to the date of event, which is defined as at least 10 points relative to baseline worsening of the GHS/QoL score or death due to any cause. If a subject had not had an event, the time to deterioration was censored at the date of the last adequate assessment. The distribution was estimated using KM method.
Time Frame: From baseline to date of at least 10 points relative to baseline worsening of the global health status score or death due to any cause, up to 2.8 years (Part 3)
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 2: Placebo + Dabrafenib 150 mg BID + Trametinib 2 mg QD
Number analyzed (Participants) | 267 | 265
Months | 19.4 [15.7 to 24.9] | 22.1 [17.5 to NA] — Not estimable (NA) due to the insufficient number of participants with events
Statistical Analysis 1: Comparison: Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD vs Part 3- Arm 2: Placebo + Dabrafenib 150 mg BID + Trametinib 2 mg QD; Test type: Superiority; p = 0.2975, Log Rank; Hazard Ratio (HR) = 1.183, 95% CI 2-sided [0.865 to 1.619]

13. Secondary Outcome: Randomized (Part 3): Change From Baseline in Function Assessment Cancer Therapy-melanoma (FACT-M) Melanoma Subscale Score
Description: The Functional Assessment of Cancer Therapy-Melanoma (FACT-M) quality of life questionnaire was composed of the FACT-General (FACT-G) plus the Melanoma Subscale and the Melanoma Surgery Subscale, which complemented the general scale with items specific to quality of life (QoL) in melanoma. The Melanoma Subscale of FACT-M included 16 questions, with response options of 0= "Not at all", 1= "a little bit", 2= "somewhat", 3= "quite a bit" and 4= "very much". The FACT-M melanoma subscale score ranged from 0 to 64, with higher scores indicating a higher quality of life in relation to melanoma. The change from baseline in melanoma subscale scores was calculated. A positive change from baseline indicated improvement.
Time Frame: From baseline to 60 days post progression, assessed up to 2.8 years (Part 3)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 2: Placebo + Dabrafenib 150 mg BID + Trametinib 2 mg QD
Number analyzed (Participants) | 177 | 190
Score on a scale
  Cycle 4 Day 1 | 0.83 (6.600) | 0.87 (6.185)
  Cycle 6 Day 1: number analyzed (Participants) | 157 | 159
  Cycle 6 Day 1 | 1.01 (7.370) | 1.18 (6.219)
  Cycle 8 Day 1: number analyzed (Participants) | 145 | 150
  Cycle 8 Day 1 | 1.14 (7.284) | 1.09 (5.742)
  Cycle 10 Day 1: number analyzed (Participants) | 133 | 125
  Cycle 10 Day 1 | 1.52 (7.314) | 0.54 (6.492)
  Cycle 12 Day 1: number analyzed (Participants) | 110 | 112
  Cycle 12 Day 1 | 1.21 (7.515) | 0.47 (5.974)
  Cycle 14 Day 1: number analyzed (Participants) | 102 | 106
  Cycle 14 Day 1 | 0.77 (7.071) | 0.65 (6.681)
  Cycle 16 Day 1: number analyzed (Participants) | 90 | 92
  Cycle 16 Day 1 | 0.93 (6.451) | 0.71 (6.374)
  Cycle 18 Day 1: number analyzed (Participants) | 88 | 86
  Cycle 18 Day 1 | 1.23 (7.095) | 0.47 (6.152)
  Cycle 20 Day 1: number analyzed (Participants) | 82 | 83
  Cycle 20 Day 1 | 1.28 (6.634) | 0.53 (5.875)
  Cycle 22 Day 1: number analyzed (Participants) | 79 | 80
  Cycle 22 Day 1 | 1.87 (6.215) | 0.79 (5.970)
  Cycle 25 Day 1: number analyzed (Participants) | 64 | 70
  Cycle 25 Day 1 | 2.73 (5.950) | 0.74 (6.792)
  Cycle 28 Day 1: number analyzed (Participants) | 50 | 56
  Cycle 28 Day 1 | 2.46 (5.195) | 0.61 (8.020)
  Cycle 31 Day 1: number analyzed (Participants) | 21 | 26
  Cycle 31 Day 1 | 3.29 (5.702) | 1.88 (6.154)
  Cycle 34 Day 1: number analyzed (Participants) | 2 | 5
  Cycle 34 Day 1 | -0.50 (2.121) | 4.60 (3.578)
  30 days post-progression: number analyzed (Participants) | 24 | 29
  30 days post-progression | 0.33 (7.620) | -1.07 (8.590)
  60 days post-progression: number analyzed (Participants) | 13 | 16
  60 days post-progression | -2.60 (5.734) | -3.06 (8.948)

14. Secondary Outcome: Randomized (Part 3): Change From Baseline in EuroQoL 5-level Instrument (EQ-5D-5L)- Visual Analog Scale (VAS) Score
Description: The EQ-5D-5L is a standardized questionnaire used to assess health-related quality of life, and it includes a Visual Analog Scale (VAS). The VAS score is obtained by asking the individual to rate their current health status on a scale from 0 to 100, where 0 represents the worst possible health state and 100 represents the best possible health state. The change from baseline in EQ-5D-5L VAS score was calculated. A positive change from baseline indicates improvement in the health status.
Time Frame: From baseline to 60 days post progression, assessed up to 2.8 years (Part 3)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 2: Placebo + Dabrafenib 150 mg BID + Trametinib 2 mg QD
Number analyzed (Participants) | 176 | 190
Score on a Scale
  Cycle 4 Day 1 | 1.85 (16.567) | 2.16 (19.733)
  Cycle 6 Day 1: number analyzed (Participants) | 156 | 158
  Cycle 6 Day 1 | 1.55 (20.751) | 3.10 (16.095)
  Cycle 8 Day 1: number analyzed (Participants) | 145 | 149
  Cycle 8 Day 1 | 0.39 (20.246) | 2.60 (15.200)
  Cycle 10 Day 1: number analyzed (Participants) | 132 | 124
  Cycle 10 Day 1 | 2.45 (19.050) | 2.52 (16.144)
  Cycle 12 Day 1: number analyzed (Participants) | 110 | 113
  Cycle 12 Day 1 | 1.88 (24.653) | 1.42 (15.695)
  Cycle 14 Day 1: number analyzed (Participants) | 102 | 107
  Cycle 14 Day 1 | 2.62 (19.455) | 1.71 (14.337)
  Cycle 16 Day 1: number analyzed (Participants) | 89 | 91
  Cycle 16 Day 1 | 1.30 (18.640) | 2.79 (16.996)
  Cycle 18 Day 1: number analyzed (Participants) | 88 | 86
  Cycle 18 Day 1 | 2.16 (20.762) | 1.91 (16.743)
  Cycle 20 Day 1: number analyzed (Participants) | 82 | 83
  Cycle 20 Day 1 | 1.34 (17.831) | 1.28 (16.108)
  Cycle 22 Day 1: number analyzed (Participants) | 79 | 80
  Cycle 22 Day 1 | 3.01 (19.102) | 1.55 (14.973)
  Cycle 25 Day 1: number analyzed (Participants) | 64 | 69
  Cycle 25 Day 1 | 4.47 (19.489) | 0.26 (14.784)
  Cycle 28 Day 1: number analyzed (Participants) | 49 | 56
  Cycle 28 Day 1 | 4.20 (17.545) | -0.39 (18.529)
  Cycle 31 Day 1: number analyzed (Participants) | 22 | 26
  Cycle 31 Day 1 | 6.45 (19.561) | -0.08 (16.747)
  Cycle 34 Day 1: number analyzed (Participants) | 2 | 5
  Cycle 34 Day 1 | -9.50 (14.849) | 5.60 (19.008)
  30 days post-progression: number analyzed (Participants) | 24 | 29
  30 days post-progression | -4.04 (22.033) | -10.24 (23.532)
  60 days post-progression: number analyzed (Participants) | 12 | 16
  60 days post-progression | -19.25 (19.923) | -8.19 (21.192)

15. Secondary Outcome: Randomized (Part 3): PFS as Per Investigator's Assessment by RECIST 1.1 by PD-L1 Expression
Description: PFS was defined as the time from the date of first dose to the date of the first documented radiological progression as per investigator's assessment using RECIST 1.1 response criteria or death due to any cause. The distribution of PFS was estimated using the KM method. If a patient had not had an event at the time of data cut-off, progression-free survival was censored at the date of last adequate tumor assessment. PFS analysis was performed by PD-L1 status (positive, negative) where a positive status was defined as having ≥ 1% expression and a negative status was defined as having < 1% expression.
Time Frame: Up to disease progression or death due to any cause, up to 2.8 years (Part 3)
Population: All participants in Part 3 to whom study treatment was assigned by randomization (regardless of whether or not treatment was administered) with an evaluable PD-L1 assessment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 2: Placebo + Dabrafenib 150 mg BID + Trametinib 2 mg QD
Number analyzed (Participants) | 236 | 241
Months
  PD-L1 negative (<1%): number analyzed (Participants) | 98 | 115
  PD-L1 negative (<1%) | 12.0 [10.1 to 15.7] | 10.3 [7.5 to 13.0]
  PD-L1 positive (>=1%): number analyzed (Participants) | 138 | 126
  PD-L1 positive (>=1%) | 26.6 [17.4 to NA] — Not estimable (NA) due to the insufficient number of participants with events | 15.4 [10.2 to 25.3]

16. Secondary Outcome: Randomized (Part 3): OS by PD-L1 Expression
Description: Overall survival was defined as the time from date of randomization to date of death due to any cause. OS analysis was performed by PD-L1 subgroup (positive, negative) where a positive status was defined as having ≥ 1% expression and a negative status was defined as having < 1% expression.
Time Frame: Up to death due to any cause, assessed up to approximately 7 years
Population: as for outcome 15
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 2: Placebo + Dabrafenib 150 mg BID + Trametinib 2 mg QD
Number analyzed (Participants) | 112 | 138
Months
  PD-L1 negative (<1%): number analyzed (Participants) | 54 | 74
  PD-L1 negative (<1%) | 41.6 [27.6 to NA] — Not estimable (NA) due to the insufficient number of participants with events | 21.0 [16.9 to 33.4]
  PD-L1 positive (>=1%): number analyzed (Participants) | 58 | 64
  PD-L1 positive (>=1%) | NA [45.4 to NA] — Not estimable (NA) due to the insufficient number of participants with events | 61.3 [41.2 to NA] — Not estimable (NA) due to the insufficient number of participants with events

17. Secondary Outcome: Spartalizumab Anti-drug Antibody (ADA) Prevalence at Baseline
Description: Spartalizumab ADA prevalence at baseline was calculated as the percentage of participants who had an spartalizumab ADA positive result at baseline.
Time Frame: Baseline
Population: Part 1 and 2: All subjects to whom study treatment was assigned and who received any study treatment with a determinant baseline immunogenicity sample and at least one determinant post-baseline immunogenicity sample. Part 3: All subjects randomized to spartalizumab with dabrafenib and trametinib with a determinant baseline immunogenicity sample and at least one determinant post-baseline immunogenicity sample. Determinant sample: sample that is neither ADA-inconclusive nor unevaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1- Safety run-in: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 2- Biomarker Cohort: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD
Number analyzed (Participants) | 9 | 26 | 244
Participants | 0 | 0 | 4

18. Secondary Outcome: Spartalizumab ADA Incidence
Description: Spartalizumab ADA incidence was calculated as the percentage of participants who were treatment-induced spartalizumab ADA positive (post-baseline ADA positive with ADA-negative sample at baseline) and treatment-boosted spartalizumab ADA positive (post-baseline ADA positive with titer that is at least the fold titer change greater than the ADA-positive baseline titer)
Time Frame: Throughout study until 150 days after the last dose of spartalizumab, up to 3.3 years (Part 1), 3 years (Part 2) and 2.8 years (Part 3).
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1- Safety run-in: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 2- Biomarker Cohort: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD
Number analyzed (Participants) | 9 | 26 | 244
Participants | 0 | 5 | 55

19. Secondary Outcome: Trough Concentration (Ctrough) for Spartalizumab
Description: Ctrough for spartalizumab refers to the serum concentration of spartalizumab immediately prior to the administration of a dose of spartalizumab on Day 1 of Cycle 2 and later cycles.
Time Frame: Pre-infusion on Day 1 of each Cycle starting from Cycle 2, up to 3.3 years (Part 1), 3 years (Part 2) and 2.8 years (Part 3). Cycle=28 days
Population: All subjects who provided at least one evaluable spartalizumab PK concentration at the specified time points.
Measure: Mean (Standard Deviation); unit: microgram (μg)/miliLiter (mL)
Arm/Group | Part 1- Safety run-in: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 2- Biomarker Cohort: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD
Number analyzed (Participants) | 5 | 17 | 138
microgram (μg)/miliLiter (mL)
  Cycle 2 | 31.9 (4.59) | 31.5 (20.3) | 28.4 (13.4)
  Cycle 3: number analyzed (Participants) | 2 | 13 | 129
  Cycle 3 | 41.1 (7.07) | 56.1 (34.2) | 43.5 (19.1)
  Cycle 4: number analyzed (Participants) | 1 | 11 | 121
  Cycle 4 | 47.8 | 46.9 (18.8) | 50.5 (24.2)
  Cycle 5: number analyzed (Participants) | 1 | 11 | 126
  Cycle 5 | 46.3 | 56.7 (19.5) | 56.4 (24.5)
  Cycle 6: number analyzed (Participants) | 5 | 9 | 119
  Cycle 6 | 53.8 (16.9) | 60.9 (23.6) | 58.8 (26.5)
  Cycle 7: number analyzed (Participants) | 4 | 8 | 119
  Cycle 7 | 56.1 (12.1) | 62.2 (33.3) | 63.7 (29.6)
  Cycle 8: number analyzed (Participants) | 2 | 7 | 104
  Cycle 8 | 57.9 (12.7) | 65.8 (32.8) | 64.1 (29.9)
  Cycle 9: number analyzed (Participants) | 5 | 6 | 88
  Cycle 9 | 60.2 (30.9) | 69.5 (25.2) | 67.8 (33.5)
  Cycle 10: number analyzed (Participants) | 2 | 4 | 87
  Cycle 10 | 62.1 (22.5) | 68.4 (33.2) | 63.8 (28.4)
  Cycle 11: number analyzed (Participants) | 2 | 7 | 91
  Cycle 11 | 66.9 (15.8) | 63.2 (35.8) | 62.1 (27.9)
  Cycle 12: number analyzed (Participants) | 5 | 5 | 85
  Cycle 12 | 67.0 (16.5) | 61.6 (29.3) | 60.7 (27.2)

20. Secondary Outcome: Pre-dose Plasma Concentration for Dabrafenib
Description: Plasma concentration of dabrafenib immediately prior to the administration of a dose of dabrafenib.
Time Frame: Pre-infusion on Day 1 of every cycle from Cycle 2 to 12, and then every 6 cycles from Cycle 18 to 36, up to 3.3 years (Part 1), 3 years (Part 2) and 2.8 years (Part 3). Cycle=28 days
Population: All subjects who provided at least one evaluable dabrafenib PK concentration at the specified time points.
Measure: Mean (Standard Deviation); unit: nanogram (ng)/ miliLiter (mL)
Arm/Group | Part 1- Safety run-in: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 2- Biomarker Cohort: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 2: Placebo + Dabrafenib 150 mg BID + Trametinib 2 mg QD
Number analyzed (Participants) | 4 | 18 | 127 | 162
nanogram (ng)/ miliLiter (mL)
  Cycle 2: number analyzed (Participants) | 3 | 18 | 125 | 162
  Cycle 2 | 33.7 (27.4) | 149 (391) | 208 (473) | 234 (475)
  Cycle 3: number analyzed (Participants) | 3 | 12 | 127 | 145
  Cycle 3 | 25.5 (10.4) | 183 (469) | 192 (607) | 135 (266)
  Cycle 4: number analyzed (Participants) | 3 | 12 | 116 | 131
  Cycle 4 | 23.0 (15.8) | 372 (811) | 169 (404) | 167 (328)
  Cycle 5: number analyzed (Participants) | 3 | 10 | 110 | 125
  Cycle 5 | 28.8 (30.6) | 152 (293) | 130 (317) | 152 (363)
  Cycle 6: number analyzed (Participants) | 3 | 10 | 110 | 113
  Cycle 6 | 15.1 (16.3) | 73.7 (131) | 198 (521) | 94.6 (186)
  Cycle 7: number analyzed (Participants) | 4 | 8 | 102 | 111
  Cycle 7 | 20.9 (13.9) | 40.0 (20.0) | 180 (510) | 121 (279)
  Cycle 8: number analyzed (Participants) | 3 | 5 | 97 | 96
  Cycle 8 | 22.9 (16.8) | 28.0 (10.4) | 173 (532) | 97.2 (177)
  Cycle 9: number analyzed (Participants) | 3 | 6 | 91 | 79
  Cycle 9 | 22.3 (7.59) | 43.3 (40.6) | 143 (394) | 133 (259)
  Cycle 10: number analyzed (Participants) | 2 | 4 | 81 | 85
  Cycle 10 | 24.5 (9.19) | 60.0 (28.3) | 167 (472) | 122 (266)
  Cycle 11: number analyzed (Participants) | 3 | 6 | 79 | 77
  Cycle 11 | 154 (250) | 33.8 (22.6) | 174 (667) | 119 (238)
  Cycle 12: number analyzed (Participants) | 3 | 4 | 75 | 67
  Cycle 12 | 10.9 (10.3) | 41.3 (37.2) | 148 (396) | 146 (295)
  Cycle 18: number analyzed (Participants) | 1 | 2 | 24 | 20
  Cycle 18 | 19.0 | 50.6 (49.7) | 180 (618) | 167 (385)
  Cycle 24: number analyzed (Participants) | 0 | 2 | 19 | 15
  Cycle 24 |  | 91.5 (98.3) | 147 (344) | 60.2 (67.9)
  Cycle 30: number analyzed (Participants) | 1 | 0 | 6 | 4
  Cycle 30 | 40.2 |  | 226 (488) | 47.6 (23.2)
  Cycle 36: number analyzed (Participants) | 1 | 0 | 0 | 0
  Cycle 36 | 47.6 |  |  |

21. Secondary Outcome: Pre-dose Plasma Concentration for Trametinib
Description: Plasma concentration of trametinib immediately prior to the administration of a dose of trametinib.
Time Frame: as for outcome 20
Population: All subjects who provided at least one evaluable trametinib PK concentration at the specified time points.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1- Safety run-in: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 2- Biomarker Cohort: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 2: Placebo + Dabrafenib 150 mg BID + Trametinib 2 mg QD
Number analyzed (Participants) | 3 | 14 | 103 | 143
ng/mL
  Cycle 2 | 11.7 (4.09) | 11.2 (3.4) | 11.5 (4.73) | 13.9 (9.36)
  Cycle 3: number analyzed (Participants) | 2 | 12 | 100 | 131
  Cycle 3 | 8.34 (0.354) | 12.2 (2.55) | 11.4 (5.98) | 12.3 (5.59)
  Cycle 4: number analyzed (Participants) | 2 | 13 | 102 | 117
  Cycle 4 | 10.7 (1.64) | 12.5 (4.84) | 11.7 (4.62) | 11.9 (5.04)
  Cycle 5: number analyzed (Participants) | 1 | 10 | 100 | 114
  Cycle 5 | 10.1 | 12.6 (5.03) | 11.3 (4.91) | 11.6 (4.49)
  Cycle 6: number analyzed (Participants) | 2 | 6 | 99 | 103
  Cycle 6 | 10.0 (1.38) | 11.8 (3.73) | 11.6 (5.12) | 10.9 (3.52)
  Cycle 7: number analyzed (Participants) | 2 | 6 | 95 | 97
  Cycle 7 | 11.6 (3.8) | 11.8 (5.24) | 12.0 (4.86) | 11.0 (4.26)
  Cycle 8: number analyzed (Participants) | 2 | 5 | 87 | 94
  Cycle 8 | 9.24 (3.06) | 10.2 (4.13) | 10.3 (3.92) | 11.3 (4.08)
  Cycle 9: number analyzed (Participants) | 2 | 6 | 78 | 75
  Cycle 9 | 8.73 (3.35) | 10.5 (4.43) | 10.9 (4.57) | 11.6 (4.22)
  Cycle 10: number analyzed (Participants) | 1 | 3 | 71 | 85
  Cycle 10 | 8.24 | 10.5 (4.02) | 10.9 (4.47) | 11.8 (4.26)
  Cycle 11: number analyzed (Participants) | 1 | 5 | 71 | 71
  Cycle 11 | 10.7 | 11.6 (4.69) | 10.3 (3.67) | 11.4 (3.57)
  Cycle 12: number analyzed (Participants) | 2 | 4 | 65 | 65
  Cycle 12 | 10.6 (3.92) | 11.0 (4.53) | 10.6 (4.31) | 11.2 (3.82)
  Cycle 18: number analyzed (Participants) | 1 | 2 | 25 | 21
  Cycle 18 | 10.1 | 13.0 (4.6) | 9.66 (3.49) | 12.1 (5.13)
  Cycle 24: number analyzed (Participants) | 0 | 2 | 17 | 12
  Cycle 24 |  | 13.4 (8.03) | 10.7 (4.89) | 10.7 (2.21)
  Cycle 30: number analyzed (Participants) | 1 | 0 | 5 | 4
  Cycle 30 | 10.8 |  | 9.34 (7.56) | 10.1 (2.76)
  Cycle 36: number analyzed (Participants) | 1 | 0 | 0 | 0
  Cycle 36 | 8.97 |  |  |

22. Secondary Outcome: Number of Participants With Dose Interruptions
Description: Number of participants with dose interruptions for spartalizumab, dabrafenib and trametinib
Time Frame: From baseline to end of treatment, assessed up to approximately 7 years
Population: All participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1- Safety run-in: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 2- Biomarker Cohort: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 2: Placebo + Dabrafenib 150 mg BID + Trametinib 2 mg QD
Number analyzed (Participants) | 9 | 27 | 267 | 264
Participants
  Spartalizumab (PDR001): With no dose interruption | 4 | 11 | 120 | 170
  Spartalizumab (PDR001): With at least one dose interruption | 5 | 16 | 147 | 94
  Dabrafenib: With no dose interruption | 0 | 2 | 29 | 74
  Dabrafenib: With at least one dose interruption | 9 | 25 | 238 | 190
  Trametinib: With no dose interruption | 0 | 1 | 29 | 64
  Trametinib: With at least one dose interruption | 9 | 26 | 238 | 200

23. Secondary Outcome: Number of Participants With Dose Reductions
Description: Number of patients with dose reductions for spartalizumab, dabrafenib and trametinib
Time Frame: From baseline to end of treatment, assessed up to approximately 7 years
Population: All participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1- Safety run-in: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 2- Biomarker Cohort: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 2: Placebo + Dabrafenib 150 mg BID + Trametinib 2 mg QD
Number analyzed (Participants) | 9 | 27 | 267 | 264
Participants
  Dabrafenib: With neither dose reduction nor interruption | 0 | 2 | 25 | 68
  Dabrafenib: With at least one dose reduction and/or interruption | 9 | 25 | 242 | 196
  Trametinib: With neither dose reduction nor interruption | 0 | 1 | 28 | 63
  Trametinib: With at least one dose reduction and/or interruption | 9 | 26 | 239 | 201

24. Secondary Outcome: Relative Dose Intensity
Description: Relative dose intensity for spartalizumab, dabrafenib and trametinib computed as the ratio (expressed as percentage) of dose intensity and planned dose intensity:
  * Spartalizumab (PDR001) = [Dose intensity (mg/4W) / planned dose intensity (mg/4W)]*100.
  * Trametinib and Dabrafenib = [Dose intensity (mg/day) / planned dose intensity (mg/day)]*100.
Time Frame: From baseline to end of treatment, assessed up to approximately 7 years
Population: All participants who received at least one dose of study treatment
Measure: Mean (Standard Deviation); unit: Percentage of planned dose intensity
Arm/Group | Part 1- Safety run-in: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 2- Biomarker Cohort: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 2: Placebo + Dabrafenib 150 mg BID + Trametinib 2 mg QD
Number analyzed (Participants) | 9 | 27 | 267 | 264
Percentage of planned dose intensity
  Spartalizumab (PDR001) | 90.7 (16.83) | 91.7 (10.41) | 94.4 (9.21) | 97.5 (5.33)
  Dabrafenib | 62.2 (26.36) | 71.3 (21.13) | 78.1 (21.21) | 89.6 (15.10)
  Trametinib | 65.9 (16.90) | 76.2 (17.19) | 79.8 (19.58) | 89.5 (14.86)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from first dose of study medication until the last dose plus 30 days safety follow-up, assessed up to approximately 86 months. Deaths were recorded from study start date until end of extended follow-up phase (end of study), assessed up to approximately 90 months.
Description: Deaths in the extended follow-up (efficacy follow-up period or survival follow-up period) were not considered adverse events. The total number at risk in the extended follow-up included patients who entered this period. All-cause Mortality was assessed for all participants enrolled in the study, while Serious and Other Adverse Events were assessed for all participants who received at least one dose of the study medication.
Groups:
- Part 1- Safety run-in: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD: Part 1- Safety run-in: PDR001 400 mg Q4W + dabrafenib 150 mg BID + trametinib 2 mg QD - Events up to 30 days safety follow-up
- Part 2- Biomarker Cohort: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD: Part 2- Biomarker cohort: PDR001 400 mg Q4W + dabrafenib 150 mg BID + trametinib 2 mg QD - Events up to 30 days safety follow-up
- Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD: Part 3- Arm 1: PDR001 400 mg Q4W + dabrafenib 150 mg BID + trametinib 2 mg QD - Events up to 30 days safety follow-up
- Part 3- Arm 2: Placebo + Dabrafenib 150 mg BID + Trametinib 2 mg QD: Part 3- Arm 2: Placebo + dabrafenib 150 mg BID + trametinib 2 mg QD - Events up to 30 days safety follow-up
- Part 1- Safety run-in: PDR001 400 mg Q4W+Dabrafenib 150 mg BID+Trametinib 2 mg QD (Extended F/Up): Part 1- Safety run-in: Spartalizumab (PDR001) 400 mg Q4W + dabrafenib 150 mg BID + trametinib 2 mg QD (Extended F/Up) - Deaths in the extended follow-up (efficacy follow-up period or survival follow-up period) were not considered adverse events.
- Part 2- Biomarker Cohort: PDR001 400 mg Q4W+Dabrafenib 150 mg BID+Trametinib 2 mg QD(Extended F/Up): Part 2- Biomarker cohort: Spartalizumab (PDR001) 400 mg Q4W + dabrafenib 150 mg BID + trametinib 2 mg QD (Extended F/Up) - Deaths in the extended follow-up (efficacy follow-up period or survival follow-up period) were not considered adverse events.
- Part 3- Arm 1: PDR001 400 mg Q4W+Dabrafenib 150 mg BID+Trametinib 2 mg QD (Extended F/Up): Part 3- Arm 1: Spartalizumab (PDR001) 400 mg Q4W + dabrafenib 150 mg BID + trametinib 2 mg QD (Extended F/Up) - Deaths in the extended follow-up (efficacy follow-up period or survival follow-up period) were not considered adverse events.
- Part 3- Arm 2: Placebo+Dabrafenib 150 mg BID+Trametinib 2 mg QD (Extended F/Up): Part 3- Arm 2: Placebo + dabrafenib 150 mg BID + trametinib 2 mg QD (Extended F/Up) - Deaths in the extended follow-up (efficacy follow-up period or survival follow-up period) were not considered adverse events.
Arm/Group | Part 1- Safety run-in: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 2- Biomarker Cohort: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 3- Arm 2: Placebo + Dabrafenib 150 mg BID + Trametinib 2 mg QD | Part 1- Safety run-in: PDR001 400 mg Q4W+Dabrafenib 150 mg BID+Trametinib 2 mg QD (Extended F/Up) | Part 2- Biomarker Cohort: PDR001 400 mg Q4W+Dabrafenib 150 mg BID+Trametinib 2 mg QD(Extended F/Up) | Part 3- Arm 1: PDR001 400 mg Q4W+Dabrafenib 150 mg BID+Trametinib 2 mg QD (Extended F/Up) | Part 3- Arm 2: Placebo+Dabrafenib 150 mg BID+Trametinib 2 mg QD (Extended F/Up)
All-Cause Mortality (participants affected / at risk) | 2/9 | 3/27 | 28/267 | 33/265 | 1/7 | 15/24 | 99/239 | 117/232
Serious Adverse Events (participants affected / at risk) | 7/9 | 18/27 | 150/267 | 123/264 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 9/9 | 27/27 | 262/267 | 250/264 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1- Safety run-in: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD (N=9) | Part 2- Biomarker Cohort: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD (N=27) | Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD (N=267) | Part 3- Arm 2: Placebo + Dabrafenib 150 mg BID + Trametinib 2 mg QD (N=264) | Part 1- Safety run-in: PDR001 400 mg Q4W+Dabrafenib 150 mg BID+Trametinib 2 mg QD (Extended F/Up) (N=0) | Part 2- Biomarker Cohort: PDR001 400 mg Q4W+Dabrafenib 150 mg BID+Trametinib 2 mg QD(Extended F/Up) (N=0) | Part 3- Arm 1: PDR001 400 mg Q4W+Dabrafenib 150 mg BID+Trametinib 2 mg QD (Extended F/Up) (N=0) | Part 3- Arm 2: Placebo+Dabrafenib 150 mg BID+Trametinib 2 mg QD (Extended F/Up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | NA | NA | NA | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 2 | 2 | NA | NA | NA | NA
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
Cardiac disorder (Cardiac disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 3 | 1 | NA | NA | NA | NA
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Hypophysitis (Endocrine disorders) | 1 | 0 | 1 | 0 | NA | NA | NA | NA
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Angle closure glaucoma (Eye disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Detachment of retinal pigment epithelium (Eye disorders) | 0 | 1 | 2 | 1 | NA | NA | NA | NA
Diplopia (Eye disorders) | 0 | 0 | 1 | 2 | NA | NA | NA | NA
Iridocyclitis (Eye disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Macular detachment (Eye disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Retinal degeneration (Eye disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Retinal detachment (Eye disorders) | 0 | 1 | 1 | 0 | NA | NA | NA | NA
Uveitis (Eye disorders) | 0 | 0 | 3 | 1 | NA | NA | NA | NA
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 5 | 1 | NA | NA | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | NA | NA | NA | NA
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Ascites (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | NA | NA | NA | NA
Autoimmune colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Colitis (Gastrointestinal disorders) | 0 | 0 | 5 | 0 | NA | NA | NA | NA
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 3 | 2 | NA | NA | NA | NA
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | NA | NA | NA | NA
Pancreatitis (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | NA | NA | NA | NA
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3 | 5 | NA | NA | NA | NA
Administration site extravasation (General disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Asthenia (General disorders) | 0 | 0 | 4 | 0 | NA | NA | NA | NA
Chills (General disorders) | 0 | 0 | 3 | 0 | NA | NA | NA | NA
Discomfort (General disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Fatigue (General disorders) | 0 | 0 | 3 | 2 | NA | NA | NA | NA
General physical health deterioration (General disorders) | 0 | 1 | 2 | 0 | NA | NA | NA | NA
Generalised oedema (General disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Influenza like illness (General disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Malaise (General disorders) | 0 | 0 | 0 | 2 | NA | NA | NA | NA
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Pain (General disorders) | 0 | 0 | 2 | 1 | NA | NA | NA | NA
Pyrexia (General disorders) | 4 | 4 | 46 | 16 | NA | NA | NA | NA
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 4 | 0 | NA | NA | NA | NA
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | NA | NA | NA | NA
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | NA | NA | NA | NA
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 2 | 0 | NA | NA | NA | NA
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Contrast media allergy (Immune system disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Sarcoidosis (Immune system disorders) | 0 | 0 | 2 | 0 | NA | NA | NA | NA
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Appendicitis perforated (Infections and infestations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Bacterial food poisoning (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Bacterial sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Biliary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Cellulitis (Infections and infestations) | 1 | 1 | 5 | 1 | NA | NA | NA | NA
Device related infection (Infections and infestations) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Empyema (Infections and infestations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Febrile infection (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | NA | NA | NA | NA
Meningitis (Infections and infestations) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Pneumonia (Infections and infestations) | 1 | 1 | 5 | 3 | NA | NA | NA | NA
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Post procedural sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Sepsis (Infections and infestations) | 0 | 0 | 5 | 3 | NA | NA | NA | NA
Septic shock (Infections and infestations) | 0 | 1 | 2 | 1 | NA | NA | NA | NA
Skin infection (Infections and infestations) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Sweating fever (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Systemic infection (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Urinary tract infection (Infections and infestations) | 0 | 0 | 3 | 0 | NA | NA | NA | NA
Urinary tract infection fungal (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Urosepsis (Infections and infestations) | 0 | 1 | 3 | 0 | NA | NA | NA | NA
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | NA | NA | NA | NA
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | NA | NA | NA | NA
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Post embolisation syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Alanine aminotransferase abnormal (Investigations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | NA | NA | NA | NA
Amylase increased (Investigations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Aspartate aminotransferase abnormal (Investigations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 2 | 0 | NA | NA | NA | NA
Blood creatinine increased (Investigations) | 0 | 0 | 4 | 0 | NA | NA | NA | NA
Body temperature increased (Investigations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
C-reactive protein increased (Investigations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Ejection fraction decreased (Investigations) | 1 | 3 | 17 | 15 | NA | NA | NA | NA
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
General physical condition abnormal (Investigations) | 0 | 1 | 2 | 1 | NA | NA | NA | NA
Hepatic enzyme increased (Investigations) | 0 | 1 | 1 | 0 | NA | NA | NA | NA
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Streptococcus test positive (Investigations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Transaminases increased (Investigations) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | NA | NA | NA | NA
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 2 | NA | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 4 | NA | NA | NA | NA
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | NA | NA | NA | NA
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | NA | NA | NA | NA
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | NA | NA | NA | NA
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2 | 3 | NA | NA | NA | NA
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 2 | NA | NA | NA | NA
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 3 | NA | NA | NA | NA
Cerebral haematoma (Nervous system disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 3 | 1 | NA | NA | NA | NA
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 3 | NA | NA | NA | NA
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | NA | NA | NA | NA
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 2 | NA | NA | NA | NA
Epilepsy (Nervous system disorders) | 0 | 0 | 2 | 2 | NA | NA | NA | NA
Headache (Nervous system disorders) | 0 | 0 | 3 | 4 | NA | NA | NA | NA
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Immune-mediated encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Intracranial tumour haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Meningism (Nervous system disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Monoparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Nerve compression (Nervous system disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Neuritis (Nervous system disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
Neurological decompensation (Nervous system disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 2 | 0 | NA | NA | NA | NA
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Polyneuropathy (Nervous system disorders) | 0 | 0 | 2 | 3 | NA | NA | NA | NA
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Seizure (Nervous system disorders) | 0 | 0 | 1 | 4 | NA | NA | NA | NA
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
Syncope (Nervous system disorders) | 0 | 0 | 2 | 0 | NA | NA | NA | NA
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 2 | NA | NA | NA | NA
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 9 | 2 | NA | NA | NA | NA
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Haematuria (Renal and urinary disorders) | 0 | 0 | 2 | 0 | NA | NA | NA | NA
Immune-mediated nephritis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Nephritis (Renal and urinary disorders) | 0 | 0 | 2 | 0 | NA | NA | NA | NA
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 2 | NA | NA | NA | NA
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 2 | 0 | NA | NA | NA | NA
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Urinary retention (Renal and urinary disorders) | 0 | 0 | 2 | 1 | NA | NA | NA | NA
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Prostatic disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Autoimmune lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | NA | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | NA | NA | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | NA | NA | NA | NA
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 9 | 2 | NA | NA | NA | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 7 | 6 | NA | NA | NA | NA
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | NA | NA | NA | NA
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | NA | NA | NA | NA
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
Aneurysm ruptured (Vascular disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Embolism (Vascular disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Haematoma (Vascular disorders) | 0 | 0 | 2 | 0 | NA | NA | NA | NA
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1- Safety run-in: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD (N=9) | Part 2- Biomarker Cohort: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD (N=27) | Part 3- Arm 1: PDR001 400 mg Q4W + Dabrafenib 150 mg BID + Trametinib 2 mg QD (N=267) | Part 3- Arm 2: Placebo + Dabrafenib 150 mg BID + Trametinib 2 mg QD (N=264) | Part 1- Safety run-in: PDR001 400 mg Q4W+Dabrafenib 150 mg BID+Trametinib 2 mg QD (Extended F/Up) (N=0) | Part 2- Biomarker Cohort: PDR001 400 mg Q4W+Dabrafenib 150 mg BID+Trametinib 2 mg QD(Extended F/Up) (N=0) | Part 3- Arm 1: PDR001 400 mg Q4W+Dabrafenib 150 mg BID+Trametinib 2 mg QD (Extended F/Up) (N=0) | Part 3- Arm 2: Placebo+Dabrafenib 150 mg BID+Trametinib 2 mg QD (Extended F/Up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 4 | 10 | 49 | 31 | NA | NA | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 2 | 1 | 23 | 14 | NA | NA | NA | NA
Lymphopenia (Blood and lymphatic system disorders) | 1 | 4 | 20 | 11 | NA | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 4 | 3 | 44 | 37 | NA | NA | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3 | 24 | 10 | NA | NA | NA | NA
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 3 | 1 | NA | NA | NA | NA
Ear congestion (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | NA | NA | NA | NA
Ear pain (Ear and labyrinth disorders) | 3 | 0 | 1 | 1 | NA | NA | NA | NA
Motion sickness (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
Hyperthyroidism (Endocrine disorders) | 2 | 0 | 18 | 5 | NA | NA | NA | NA
Hypophysitis (Endocrine disorders) | 1 | 0 | 1 | 0 | NA | NA | NA | NA
Hypothyroidism (Endocrine disorders) | 4 | 1 | 20 | 17 | NA | NA | NA | NA
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
Thyroiditis (Endocrine disorders) | 1 | 1 | 3 | 0 | NA | NA | NA | NA
Dry eye (Eye disorders) | 0 | 9 | 5 | 9 | NA | NA | NA | NA
Iridocyclitis (Eye disorders) | 1 | 0 | 3 | 3 | NA | NA | NA | NA
Myopia (Eye disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
Ocular discomfort (Eye disorders) | 0 | 2 | 1 | 0 | NA | NA | NA | NA
Papilloedema (Eye disorders) | 1 | 1 | 2 | 1 | NA | NA | NA | NA
Periorbital oedema (Eye disorders) | 1 | 0 | 4 | 1 | NA | NA | NA | NA
Photophobia (Eye disorders) | 1 | 0 | 6 | 3 | NA | NA | NA | NA
Retinal haemorrhage (Eye disorders) | 1 | 0 | 1 | 0 | NA | NA | NA | NA
Retinopathy (Eye disorders) | 1 | 1 | 0 | 0 | NA | NA | NA | NA
Uveitis (Eye disorders) | 1 | 3 | 7 | 4 | NA | NA | NA | NA
Vision blurred (Eye disorders) | 0 | 2 | 9 | 13 | NA | NA | NA | NA
Visual impairment (Eye disorders) | 0 | 2 | 10 | 6 | NA | NA | NA | NA
Vitreal cells (Eye disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 2 | 5 | NA | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 1 | 5 | 29 | 26 | NA | NA | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 26 | 17 | NA | NA | NA | NA
Cheilitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | NA | NA | NA | NA
Constipation (Gastrointestinal disorders) | 1 | 7 | 40 | 40 | NA | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 4 | 9 | 98 | 70 | NA | NA | NA | NA
Dry mouth (Gastrointestinal disorders) | 1 | 6 | 22 | 13 | NA | NA | NA | NA
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 18 | 13 | NA | NA | NA | NA
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 9 | 6 | NA | NA | NA | NA
Glossitis (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | NA | NA | NA | NA
Nausea (Gastrointestinal disorders) | 1 | 8 | 90 | 78 | NA | NA | NA | NA
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 4 | 4 | NA | NA | NA | NA
Trichoglossia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 4 | 10 | 69 | 50 | NA | NA | NA | NA
Asthenia (General disorders) | 1 | 11 | 73 | 55 | NA | NA | NA | NA
Axillary pain (General disorders) | 0 | 2 | 4 | 3 | NA | NA | NA | NA
Chills (General disorders) | 8 | 9 | 86 | 63 | NA | NA | NA | NA
Face oedema (General disorders) | 1 | 0 | 8 | 2 | NA | NA | NA | NA
Fatigue (General disorders) | 7 | 11 | 71 | 69 | NA | NA | NA | NA
Influenza like illness (General disorders) | 4 | 4 | 28 | 15 | NA | NA | NA | NA
Non-cardiac chest pain (General disorders) | 2 | 1 | 5 | 1 | NA | NA | NA | NA
Oedema (General disorders) | 0 | 2 | 3 | 7 | NA | NA | NA | NA
Oedema due to cardiac disease (General disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
Oedema peripheral (General disorders) | 1 | 2 | 30 | 28 | NA | NA | NA | NA
Pain (General disorders) | 1 | 5 | 7 | 10 | NA | NA | NA | NA
Pyrexia (General disorders) | 9 | 23 | 189 | 145 | NA | NA | NA | NA
Xerosis (General disorders) | 0 | 2 | 3 | 2 | NA | NA | NA | NA
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 2 | 5 | 7 | NA | NA | NA | NA
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | NA | NA | NA | NA
Hepatitis (Hepatobiliary disorders) | 2 | 1 | 5 | 3 | NA | NA | NA | NA
Hypertransaminasaemia (Hepatobiliary disorders) | 2 | 0 | 6 | 4 | NA | NA | NA | NA
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 | 1 | 1 | 0 | NA | NA | NA | NA
Cytokine release syndrome (Immune system disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
Sarcoidosis (Immune system disorders) | 1 | 1 | 5 | 2 | NA | NA | NA | NA
Bronchitis (Infections and infestations) | 0 | 1 | 20 | 5 | NA | NA | NA | NA
COVID-19 (Infections and infestations) | 0 | 0 | 18 | 13 | NA | NA | NA | NA
Candida infection (Infections and infestations) | 1 | 0 | 0 | 2 | NA | NA | NA | NA
Cellulitis (Infections and infestations) | 1 | 2 | 6 | 2 | NA | NA | NA | NA
Conjunctivitis (Infections and infestations) | 2 | 3 | 14 | 9 | NA | NA | NA | NA
Folliculitis (Infections and infestations) | 3 | 1 | 14 | 8 | NA | NA | NA | NA
Fungal skin infection (Infections and infestations) | 1 | 0 | 2 | 1 | NA | NA | NA | NA
Furuncle (Infections and infestations) | 1 | 1 | 0 | 3 | NA | NA | NA | NA
Gastrointestinal viral infection (Infections and infestations) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Nasopharyngitis (Infections and infestations) | 2 | 3 | 28 | 32 | NA | NA | NA | NA
Oral candidiasis (Infections and infestations) | 1 | 2 | 2 | 2 | NA | NA | NA | NA
Oral herpes (Infections and infestations) | 1 | 1 | 8 | 4 | NA | NA | NA | NA
Otitis media (Infections and infestations) | 1 | 0 | 1 | 1 | NA | NA | NA | NA
Otitis media chronic (Infections and infestations) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
Paronychia (Infections and infestations) | 1 | 0 | 4 | 3 | NA | NA | NA | NA
Pneumonia (Infections and infestations) | 1 | 2 | 9 | 9 | NA | NA | NA | NA
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Rhinitis (Infections and infestations) | 1 | 1 | 18 | 10 | NA | NA | NA | NA
Sinusitis (Infections and infestations) | 1 | 2 | 12 | 2 | NA | NA | NA | NA
Tonsillitis (Infections and infestations) | 1 | 0 | 3 | 2 | NA | NA | NA | NA
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 17 | 9 | NA | NA | NA | NA
Urinary tract infection (Infections and infestations) | 0 | 5 | 26 | 25 | NA | NA | NA | NA
Viral infection (Infections and infestations) | 1 | 1 | 4 | 5 | NA | NA | NA | NA
Viral pharyngitis (Infections and infestations) | 2 | 0 | 0 | 0 | NA | NA | NA | NA
Viral rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 2 | 2 | NA | NA | NA | NA
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 2 | NA | NA | NA | NA
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 0 | NA | NA | NA | NA
Radiation skin injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 3 | 7 | 67 | 41 | NA | NA | NA | NA
Amylase increased (Investigations) | 4 | 4 | 46 | 22 | NA | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 2 | 5 | 76 | 53 | NA | NA | NA | NA
Blood albumin decreased (Investigations) | 1 | 0 | 4 | 1 | NA | NA | NA | NA
Blood alkaline phosphatase increased (Investigations) | 2 | 4 | 33 | 28 | NA | NA | NA | NA
Blood cholesterol increased (Investigations) | 1 | 3 | 12 | 11 | NA | NA | NA | NA
Blood creatine phosphokinase increased (Investigations) | 3 | 9 | 75 | 72 | NA | NA | NA | NA
Blood creatinine increased (Investigations) | 2 | 2 | 24 | 9 | NA | NA | NA | NA
Blood lactate dehydrogenase increased (Investigations) | 1 | 1 | 27 | 21 | NA | NA | NA | NA
Blood sodium decreased (Investigations) | 1 | 0 | 1 | 2 | NA | NA | NA | NA
Blood testosterone decreased (Investigations) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 0 | 5 | 2 | NA | NA | NA | NA
Blood triglycerides increased (Investigations) | 1 | 0 | 3 | 2 | NA | NA | NA | NA
C-reactive protein increased (Investigations) | 2 | 2 | 12 | 11 | NA | NA | NA | NA
Ejection fraction decreased (Investigations) | 1 | 2 | 18 | 21 | NA | NA | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 2 | 3 | 17 | 20 | NA | NA | NA | NA
Globulins increased (Investigations) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
Hepatic enzyme increased (Investigations) | 0 | 2 | 5 | 5 | NA | NA | NA | NA
Lipase increased (Investigations) | 5 | 5 | 66 | 38 | NA | NA | NA | NA
Lymphocyte count decreased (Investigations) | 0 | 2 | 5 | 5 | NA | NA | NA | NA
Myoglobin blood increased (Investigations) | 1 | 0 | 2 | 0 | NA | NA | NA | NA
Neutrophil count decreased (Investigations) | 2 | 3 | 8 | 11 | NA | NA | NA | NA
Transaminases increased (Investigations) | 0 | 2 | 9 | 6 | NA | NA | NA | NA
Weight decreased (Investigations) | 0 | 4 | 17 | 11 | NA | NA | NA | NA
White blood cell count decreased (Investigations) | 1 | 2 | 9 | 6 | NA | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 2 | 7 | 33 | 27 | NA | NA | NA | NA
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 3 | 3 | NA | NA | NA | NA
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 1 | 8 | 4 | NA | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 37 | 24 | NA | NA | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 3 | 4 | NA | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 15 | 6 | NA | NA | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2 | 17 | 4 | NA | NA | NA | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 4 | 14 | 16 | NA | NA | NA | NA
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | NA | NA | NA | NA
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1 | 5 | NA | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 15 | 87 | 80 | NA | NA | NA | NA
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 6 | 4 | NA | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 5 | 33 | 37 | NA | NA | NA | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 2 | NA | NA | NA | NA
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 7 | 1 | NA | NA | NA | NA
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 2 | 6 | 5 | NA | NA | NA | NA
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0 | NA | NA | NA | NA
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 32 | 28 | NA | NA | NA | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 8 | 4 | NA | NA | NA | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 5 | 3 | NA | NA | NA | NA
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3 | 8 | NA | NA | NA | NA
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 5 | NA | NA | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 8 | 43 | 37 | NA | NA | NA | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 7 | 9 | NA | NA | NA | NA
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1 | NA | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 6 | 31 | 23 | NA | NA | NA | NA
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | NA | NA | NA | NA
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2 | 9 | NA | NA | NA | NA
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Anosmia (Nervous system disorders) | 2 | 0 | 0 | 1 | NA | NA | NA | NA
Aphasia (Nervous system disorders) | 1 | 0 | 4 | 2 | NA | NA | NA | NA
Dizziness (Nervous system disorders) | 2 | 1 | 21 | 23 | NA | NA | NA | NA
Dizziness postural (Nervous system disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
Dysaesthesia (Nervous system disorders) | 0 | 3 | 2 | 2 | NA | NA | NA | NA
Dysgeusia (Nervous system disorders) | 0 | 3 | 13 | 6 | NA | NA | NA | NA
Headache (Nervous system disorders) | 5 | 8 | 80 | 74 | NA | NA | NA | NA
Memory impairment (Nervous system disorders) | 1 | 0 | 1 | 2 | NA | NA | NA | NA
Migraine (Nervous system disorders) | 1 | 0 | 2 | 2 | NA | NA | NA | NA
Paraesthesia (Nervous system disorders) | 0 | 5 | 14 | 14 | NA | NA | NA | NA
Peroneal nerve palsy (Nervous system disorders) | 0 | 2 | 1 | 0 | NA | NA | NA | NA
Syncope (Nervous system disorders) | 0 | 4 | 2 | 3 | NA | NA | NA | NA
Anxiety (Psychiatric disorders) | 0 | 1 | 12 | 16 | NA | NA | NA | NA
Bradyphrenia (Psychiatric disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
Disorientation (Psychiatric disorders) | 1 | 0 | 1 | 0 | NA | NA | NA | NA
Insomnia (Psychiatric disorders) | 1 | 1 | 22 | 18 | NA | NA | NA | NA
Acute kidney injury (Renal and urinary disorders) | 1 | 2 | 6 | 1 | NA | NA | NA | NA
Dysuria (Renal and urinary disorders) | 0 | 1 | 14 | 8 | NA | NA | NA | NA
Haematuria (Renal and urinary disorders) | 1 | 0 | 8 | 9 | NA | NA | NA | NA
Nocturia (Renal and urinary disorders) | 0 | 2 | 0 | 1 | NA | NA | NA | NA
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 2 | NA | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 12 | 63 | 49 | NA | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 37 | 30 | NA | NA | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 17 | 8 | NA | NA | NA | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 10 | 11 | NA | NA | NA | NA
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 28 | 4 | NA | NA | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 12 | 6 | NA | NA | NA | NA
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 10 | 5 | NA | NA | NA | NA
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | NA | NA | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 17 | 9 | NA | NA | NA | NA
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 | 2 | 13 | 14 | NA | NA | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 4 | 14 | 15 | NA | NA | NA | NA
Eczema (Skin and subcutaneous tissue disorders) | 1 | 2 | 9 | 16 | NA | NA | NA | NA
Erythema (Skin and subcutaneous tissue disorders) | 0 | 3 | 27 | 11 | NA | NA | NA | NA
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 1 | 14 | 9 | NA | NA | NA | NA
Granuloma annulare (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 1 | 7 | 14 | NA | NA | NA | NA
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 5 | 1 | NA | NA | NA | NA
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 1 | NA | NA | NA | NA
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 4 | 10 | 11 | NA | NA | NA | NA
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2 | NA | NA | NA | NA
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 2 | 9 | 8 | NA | NA | NA | NA
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 1 | 9 | 3 | NA | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 8 | 51 | 22 | NA | NA | NA | NA
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1 | NA | NA | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 4 | 13 | 76 | 68 | NA | NA | NA | NA
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 1 | 5 | 1 | NA | NA | NA | NA
Rash macular (Skin and subcutaneous tissue disorders) | 2 | 2 | 2 | 3 | NA | NA | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 3 | 16 | 6 | NA | NA | NA | NA
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 2 | 7 | 1 | NA | NA | NA | NA
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 4 | NA | NA | NA | NA
Sensitive skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | NA | NA | NA | NA
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 6 | 7 | NA | NA | NA | NA
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 2 | 21 | 3 | NA | NA | NA | NA
Hot flush (Vascular disorders) | 0 | 3 | 5 | 4 | NA | NA | NA | NA
Hypertension (Vascular disorders) | 0 | 2 | 20 | 34 | NA | NA | NA | NA
Hypotension (Vascular disorders) | 2 | 1 | 10 | 7 | NA | NA | NA | NA
Lymphoedema (Vascular disorders) | 1 | 3 | 7 | 4 | NA | NA | NA | NA
Orthostatic hypotension (Vascular disorders) | 0 | 2 | 0 | 3 | NA | NA | NA | NA
Superficial vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-01-27): https://cdn.clinicaltrials.gov/large-docs/92/NCT02967692/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT02967692/SAP_002.pdf